CLINICAL TRIAL: NCT00953979
Title: A Clinical Trial About the Efficacy and Safety of Kunxian Capsule in Treatment Patients With Early Ankylosing Spondylitis: a 12-week, Multi-center, Randomized, Double-blind, Active Drug and Placebo Compared Clinical Trial
Brief Title: Efficacy and Safety of Kunxian Capsule in Treatment Patients With Early Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gu Jieruo (Other)
Collaborators: China-Japan Friendship Hospital (Other); Dongguan People's Hospital (Other Government); Zhujiang Hospital (Other); Huashan Hospital (Other)
Responsible Party: Sponsor-Investigator, Gu Jieruo, Department of Rheumatology, the Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-2
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Ankylosing Spondylitis; Treatment
Keywords: ankylosing spondylitis; treatment; Sulfasalazine; kunxian capsule
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — kunxian

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulfasalazine (Active Comparator): Sulfasalazine is a drug in treatment RA, AS and ulcerative colonitis. In this study, Sulfasalazine is used to act as an active comparator to access the efficacy of kunxian capsule.
  Interventions: Drug: kunxian capsule
- placebo (Placebo Comparator): The placebo capsule was used to be a comparator of kunxian capsule
  Interventions: Drug: kunxian capsule

INTERVENTIONS:
Drug: kunxian capsule — The main element of kunxian capsule is Tripterygium. Patients should take 2 tablets per time and 3 times per day for 12 weeks.

SUMMARY:
This is a prospective randomized controlled study to evaluated the efficacy and safety of kunxian capsule in treating of patients with early ankylosing spondylitis (AS). The major outcome index is proportion of patients achieving ASAS20 response at week12, and minor outcome indexes include ASAS50 and ASAS70, BASDAI20,BASDAI50 and BASDAI70. The adverse events at any time were recorded to evaluate the safety.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 65 years old, having signed the informed consent;
* fulfill the ESSG criteria for diagnosis of SpA; not fulfill the 1984 modified NewYork criteria for AS;
* BASDAI score more than 4;
* stop taking DMARDs for at least 4 weeks;
* NSAIDs dosage has been stable for at least 4 weeks;

Exclusion Criteria:

* Intra-articular injection of cortisone within 3 months.
* History of heart failure, multiple sclerosis, COPD, lymphoma or other tumors;
* Accompanied by fibromyalgia or other rheumatic diseases;
* Female of pregnancy or breast feeding;
* History of mental disease and poor compliance.
* History of drug abuse or alcoholism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
proportion of patients achieving ASAS20 response | 12th week

SECONDARY OUTCOMES:
proportion of patients achieving BASDAI20/50/70 response | 12th week

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, M.D., Principal Investigator — Rheumatology Department, Third Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Rheumatology Department, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li Q, Li L, Bi L, Xiao C, Lin Z, Cao S, Liao Z, Gu J. Kunxian capsules in the treatment of patients with ankylosing spondylitis: a randomized placebo-controlled clinical trial. Trials. 2016 Jul 22;17(1):337. doi: 10.1186/s13063-016-1438-6. PMID 27449221